CLINICAL TRIAL: NCT05624411
Title: Clinical Outcomes of Post-placental Insertion of Cupper T380A and Multiload 375 Contraceptive Devices During Cesarean Section
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mahmoud Ahmed Abdelmawgoud, principal investigator, Sohag University
Other Study IDs: soh-Med-22-11-03
Record Dates: First submitted 2022-10-21; First posted 2022-11-22 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: IUD (Intrauterine Device) Malposition; IUD; Complications, Infection or Inflammation
Keywords: postplacental IUD; IUD; Cupper T380A IUD; Multiload 375 IUD; iud expulsion
MeSH Terms: conditions — Infections; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- A: post-placental insertion of CU T380A IUD during CS
  Interventions: Device: CU T380A IUD
- B: post-placental insertion of multiload 375 IUD during CS
  Interventions: Device: multiload 375 IUD

INTERVENTIONS:
Device: CU T380A IUD — post-placental insertion of intrauterine contraceptive device
  Other Names: CU T380A
  Groups: A
Device: multiload 375 IUD — post-placental insertion of intrauterine contraceptive device
  Other Names: multiload 375
  Groups: B

SUMMARY:
Clinical outcomes of post-placental insertion of Cupper T380A and Multiload 375 contraceptive devices during cesarean section

DETAILED DESCRIPTION:
An intrauterine device (IUD) is considered one of the most effective, highly convenient and cheap methods of contraception[1]. IUD has been endorsed as a first-line contraceptive choice by the American College of Obstetricians and Gynecologists [2]. However, many complications have been reported with its use, such as irregular bleeding, expulsion, pelvic pain, and unexpected pregnancy.

Furthermore, extrauterine migration of IUD may result in damage to adjacent organs, bowel injury or even death [3]. Well-designed studies have elucidated that uterine perforation is expected in 0.2 to 3.6 per 1000 IUD insertions [4]. In addition, some case reports have shown IUD displacement into the sigmoid colon and lower urinary tract [5-8].

Nearly, fifty percent of malpositioned IUDs are asymptomatic and usually undetected for many years. Taking into consideration the possible risk of extrauterine migration and its dangerous sequelas, follow-up examinations are advised for all women after IUD insertion [9].

One of the safe, trusted and most convenient strategies to avoid new unwanted pregnancies is immediate postpartum IUD placement, within 10 minutes of delivery of the placenta [10]. However, expulsion rates are higher after immediate postpartum IUD insertions in comparison to delayed postpartum insertions (4-6 weeks postpartum)[11-13] Ultrasonographic assessment is considered the standard tool for confirming the position of an IUD.

2) Aim of the study The aim of the current study is to compare two types of intrauterine devices, namely Cu T380A IUD and Multiload 375 IUD, inserted immediately post placental, as regard to expulsion rates, safety, efficacy, side effects, and complications.

3) Subjects and Methods

1) Study type: A randomized comparative clinical trial 4) Methods: This study is a clinical trial that will include all patients fulfilling the eligibility criteria and presented to the emergency unit of the department of Obstetrics and Gynecology at Sohag University hospital (Egyptian tertiary referral hospital) who are requesting immediate postpartum contraception between November 2022 and September 2023. The attending physician will explain the nature of the study and all patients included will be asked to sign an informed consent. Participants were randomly allocated through a computer-generated list into two groups. In the first group Cu-T380A (Pregna International Ltd) will be inserted while in the second group Multiload 375 (Pregna International Ltd, Mumbai, India) will be inserted, Researchers and participants will not be masked to the type of IUCD inserted.

IUCDs will be inserted high at the fundus through the lower uterine segment incision immediately after delivery of the placenta using the cylinder provided within the sterile packaging; the IUCD pushing rod will not be used. Before placement in the uterine cavity, both IUCD strings were lengthened using 10 cm of Vicryl sutures (polyglactin 910) number 0 which will then threaded through the cylinder to appear at the other end. Following insertion adjacent to the fundus, the cylinder will be gradually moved downwards across the threads, passed through the cervix, and removed vaginally after delivery [14], This technique ensures that the threads are located within the vagina immediately after the operation and prevents their entanglement within the cervical canal or uterine cavity[14]. The uterine incision will then be closed in two layers.

Transabdominal US will be done to all patients before discharge to ensure adequate position of the IUD and then Women will be requested to attend follow-up appointment at 6 weeks after delivery, gynecological examination in addition to transvaginal sonography will be done to measure top-fundal distance that reflects the position of the IUD. The participants were instructed to report the pattern of bleeding during the puerperium, the number of sanitary pads used per day, the presence of blood clots, missed periods, fever, or vaginal discharge. They were shown how to find the threads and informed to urgently seek medical care if they could not feel the threads. During the puerperium, the Vicryl suture knot appeared below the cervix; the threads were shortened to a length of 2 cm from the cervix. Transabdominal and transvaginal 2D ultrasonography will be used to evaluate IUCD position in each visit. Complete expulsion was recorded when the longitudinal arm of the IUCD was partially or totally inside the cervix or vagina. Partial expulsion or displacement was recorded when the IUCD was more than 10 mm away from the fundus but still totally within the uterine cavity [15]. Women with severe PID who did not respond to treatment and/or had severe menorrhagia were candidates for IUCD discontinuation and were prescribed another contraception method if required.

5) Statistical analysis: Data will be expressed as mean ± standard deviation (SD), unless stated otherwise. Chi-squared test will be used to compare categorical variables and Student's t-test to compare continuous variables. A p-value of <0.05 will be considered statistically significant. STATA v14 (StataCorp. 2015. Stata Statistical Software: Release 14. College Station, TX: StataCorp LP) and MedCalc programs and will be used for data analysis.

6) Study results and impact: The current study may prove or disprove the benefits versus the risks of intrapartum insertion of different types of IUCDs.

ELIGIBILITY:
Inclusion Criteria:

-(1) All patients admitted for delivery at our department who requested postpartum contraception, were invited to participate in the study.

(2) Age (18-45)

Exclusion Criteria:

* (1) Intrauterine infection at time of delivery (chorioamnionitis) (2) postpartum hemorrhage (3) Uterine anomalies (distorted uterine cavity) (4) History of previous IUD expulsion (5) Anemic patients with hemoglobin< 10gm/dl (6) pre-labor rupture of membranes for more than 18 hours (7) Placenta previa.

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Study Population: All patients admitted for delivery at obstetric and gynecology emergency unit of sohag university hospital which is a tertiary center at sohag city in egypt who requested postpartum contraception, were invited to participate in the study
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-10-22 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
The expulsion rate of Multiload IUCD versus CopperT380A after post-placental insertion | 6 weeks
  The expulsion rate of Multiload IUCD versus CopperT380A after post-placental insertion

SECONDARY OUTCOMES:
Uterine bleeding | 6 weeks
  number of bleeding days
Uterine bleeding | 6 weeks
  pattern of bleeding
Uterine bleeding | 6 weeks
  presence of blood clots
PID | 6 weeks
  pesence of fever or vaginal discharge
perforation | 6 weeks
  presence of abdominal pain
pregnancy on top of IUCD | 6 weeks
  missed periods , or pregnancy

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Egypt

REFERENCES:
- [Background] Bilian X. Chinese experience with intrauterine devices. Contraception. 2007 Jun;75(6 Suppl):S31-4. doi: 10.1016/j.contraception.2006.12.007. Epub 2007 Feb 16. PMID 17531613
- [Background] Hillard PJ. Practical tips for intrauterine devices use in adolescents. J Adolesc Health. 2013 Apr;52(4 Suppl):S40-6. doi: 10.1016/j.jadohealth.2012.09.023. PMID 23535056
- [Background] Behtash N, Akhavan S, Mokhtar S. Pelvic mass due to transmigrated IUD. Acta Med Iran. 2010 Mar-Apr;48(2):125-6. PMID 21133007
- [Background] Vasquez P, Schreiber CA. The missing IUD. Contraception. 2010 Aug;82(2):126-8. doi: 10.1016/j.contraception.2010.02.019. Epub 2010 Apr 2. No abstract available. PMID 20654751
- [Background] Ko PC, Lin YH, Lo TS. Intrauterine contraceptive device migration to the lower urinary tract: report of 2 cases. J Minim Invasive Gynecol. 2011 Sep-Oct;18(5):668-70. doi: 10.1016/j.jmig.2011.05.010. PMID 21872173
- [Background] Kus E, Swierczewski A, Pasinski J, Estemberg D, Brzozowska M, Kowalska-Koprek U, Berner-Trabska M, Karowicz-Bilinska A. [Intrauterine contraceptive device in an appendix--a case report]. Ginekol Pol. 2012 Feb;83(2):132-5. Polish. PMID 22568359
- [Background] Taras AR, Kaufman JA. Laparoscopic retrieval of intrauterine device perforating the sigmoid colon. JSLS. 2010 Jul-Sep;14(3):453-5. doi: 10.4293/108680810X12924466006684. PMID 21333209
- [Background] Vilallonga R, Rodriguez N, Vilchez M, Armengol M. Translocation of an intrauterine contraceptive device: incidental finding in the rectosigmoid colon. Obstet Gynecol Int. 2010;2010:404160. doi: 10.1155/2010/404160. Epub 2010 Jun 9. PMID 20613996
- [Background] Koltan SO, Tamay AG, Yildirim Y. Chronic cervical perforation by an intrauterine device. J Chin Med Assoc. 2010 Jun;73(6):325-6. doi: 10.1016/S1726-4901(10)70069-1. PMID 20603091
- [Background] American College of Obstetricians and Gynecologists' Committee on Obstetric Practice. Committee Opinion No. 670: Immediate Postpartum Long-Acting Reversible Contraception. Obstet Gynecol. 2016 Aug;128(2):e32-7. doi: 10.1097/AOG.0000000000001587. PMID 27454734
- [Background] Whitaker AK, Chen BA. Society of Family Planning Guidelines: Postplacental insertion of intrauterine devices. Contraception. 2018 Jan;97(1):2-13. doi: 10.1016/j.contraception.2017.09.014. Epub 2017 Oct 5. PMID 28987293
- [Background] Lopez LM, Bernholc A, Hubacher D, Stuart G, Van Vliet HA. Immediate postpartum insertion of intrauterine device for contraception. Cochrane Database Syst Rev. 2015 Jun 26;2015(6):CD003036. doi: 10.1002/14651858.CD003036.pub3. PMID 26115018
- [Background] Averbach SH, Ermias Y, Jeng G, Curtis KM, Whiteman MK, Berry-Bibee E, Jamieson DJ, Marchbanks PA, Tepper NK, Jatlaoui TC. Expulsion of intrauterine devices after postpartum placement by timing of placement, delivery type, and intrauterine device type: a systematic review and meta-analysis. Am J Obstet Gynecol. 2020 Aug;223(2):177-188. doi: 10.1016/j.ajog.2020.02.045. Epub 2020 Mar 3. PMID 32142826
- [Background] Nelson AL, Chen S, Eden R. Intraoperative placement of the Copper T-380 intrauterine devices in women undergoing elective cesarean delivery: a pilot study. Contraception. 2009 Jul;80(1):81-3. doi: 10.1016/j.contraception.2009.01.014. Epub 2009 Mar 4. PMID 19501220
- [Background] Mosley FR, Shahi N, Kurer MA. Elective surgical removal of migrated intrauterine contraceptive devices from within the peritoneal cavity: a comparison between open and laparoscopic removal. JSLS. 2012 Apr-Jun;16(2):236-41. doi: 10.4293/108680812x13427982377265. PMID 23477171